CLINICAL TRIAL: NCT04197401
Title: Screening & Health Education in Barbershop Centers for Hypertension
Acronym: SALOON-HTN
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Société Tunisienne de Cardiologie & de Chirurgie Cardiovasculaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-007-SALOONHTN
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Hypertension
Keywords: Barbershop; Screening; Health Education; Cardiology; DACIMA Clinical Suite
MeSH Terms: conditions — Hypertension; Health Education

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SALOON-HTN is a cross-sectional, descriptive, non-interventional, multicenter survey aiming to screen high blood pressure by measuring blood pressure in barbershops.

DETAILED DESCRIPTION:
The survey is a screening project for hypertension, which will enroll subjects at the barbershops. The Metline Township (located at Bizerte Town, in the north of Tunisia) will be the geographical area of population enrollment. Barbershops hairdressers will be trained by a medical staff to measure the blood pressure by an ambulatory device.

All subjects willing to participate in the survey will be asked to measure their blood pressure by after at least 5 minutes rest. Three measures will be performed by the Hairdressers, with an interval of 3 minutes between each measure. The mean of the last two measures will be considered. If the mean blood pressure level exceeds 135/85 mmHg the subject will be sent to a physician of his choice.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Informed Consent to participate in the screening study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population to enroll is represented by all men and women who are willing to screen their blood pressure level at the barbershops of Metline Township (located at Bizerte town, in the North of Tunisia).
Sampling Method: Non-Probability Sample
Enrollment: 1536 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Hypertension frequency | at inclusion
  Number of subjects with systolic blood pressure above 135 mmHg and/or diastolic blood pressure above 85 mmHg
Controlled Hypertensive patients | at inclusion
  Number of subjects with known hypertension having systolic blood pressure below 135 mmHg and diastolic blood pressure below 85 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Faouzi Addad, MD, Study Chair — Société Tunisienne de Cardiologie & de Chirurgie Cardiovasculaire
Locations (1):
- Barbershops (N = 27), Al Matlīn, Bizerte Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Screening and health education in barbershop centers for hypertension (SALOON-HTN) : ESC Congress 2020 — https://esc365.escardio.org/Congress/218621-screening-and-health-education-in-barbershop-centers-for-hypertension-saloon-htn?_ga=2.65453036.393061635.1601766393-1132881307.1601766393#abstract